CLINICAL TRIAL: NCT01038596
Title: Proliferation and Osteogenic Differentiation of Bone Marrow-derived Mesenchymal Stromal Cells From Osteoarthritic Versus Healthy Donors
Brief Title: Mesenchymal Stromal Cells and Osteoarthritis
Status: Completed | Type: Observational
Sponsor: Technische Universität Dresden (Other)
Collaborators: German Federal Ministry of Education and Research (Other Government)
Responsible Party: Sponsor
Other Study IDs: HipMSC-Osteoarthritis
Record Dates: First submitted 2009-12-23; First posted 2009-12-24 (Estimated); Last update posted 2017-04-14 (Actual); Status verified 2017-04

CONDITIONS: Osteoarthritis
Keywords: osteoarthritis, mesenchymal stromal cells, proliferation
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — bone marrow aspirates
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- osteoarthritic donors: pelvic compartment advanced-stage (Kellgren and Lawrence grade 3 or 4) osteoarthritic donors
- healthy donors: age-matched healthy donors

SUMMARY:
Osteoarthritis (OA) is one of the most frequent musculoskeletal disorders and represents the main indication for total joint arthroplasty. Multipotent mesenchymal stromal cells (MSCs) can be easily isolated and culture expanded from bone marrow aspirates and provide an excellent source of progenitor cells for cell-based regeneration strategies due to their ex vivo differentiation and proliferation capacity. Although there are hints that MSCs derived from OA patients may exhibit altered function the role of MSCs with respect to disease development and progression of OA is not clearly understood to date. To assess whether advanced-stage OA affects MSCs' suitability for musculoskeletal regenerative therapy, in the present study, we compare proliferation and differentiation potential of MSCs from osteoarthritic versus healthy donors.

DETAILED DESCRIPTION:
Clinical data (range of motion of lower limb joints, sociodemographic score dataset, WOMAC score, EQ-5D score, Harris Hip Score, radiological evaluation (OA group only), routine laboratory parameters, and bone metabolism parameters)

Osteogenic, chondrogenic, and adipogenic differentiation is proofed qualitatively by cell staining

osteogenic, chondrogenic and adipogenic marker gene expression analysis using quantitative real-time RT-PCR

cell-specific alkaline phosphatase (ALP) activity assay

large-scale gene expression profile

Fluorescence-activated cell sorting (FACS)- CD44, CD105 (SH2; endoglin), CD106 (vascular cell adhesion molecule; VCAM-1), CD166, CD29, CD73 (SH3 and SH4), CD90 (Thy-1), CD117, STRO-1 and Sca-1 [%]

ELIGIBILITY:
Inclusion Criteria:

* indication for hip THR
* primary osteoarthritis of the hip
* Patient's consent

Exclusion Criteria:

* secondary osteoarthritis of the hip
* Any malignancies
* infectious disease
* rheumatic disease
* osteoporosis
* Any additional serious disease complicating the participation in this study

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: pelvic compartment advanced-stage (Kellgren and Lawrence grade 3 or 4, mean 67±6 years) osteoarthritic and age-matched healthy donors
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2009-01; Primary Completion 2016-06 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Global Gene expression profile of bone marrow-derived mesenchymal stromal cells from osteoarthritic versus healthy donors | after msc isolation

SECONDARY OUTCOMES:
Flow cytometric analysis of cell surface antigens, Alkaline phosphatase activity, DNA content as measure for cellular proliferation | variable 2 days up to 21 days after msc cultivation

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Dresden, Orthopaedic Department, Dresden, Germany